CLINICAL TRIAL: NCT04985955
Title: A Phase 1, Single Center, Randomized, Controlled Platform Study Validating the Use of Candin as a Challenge Agent in Healthy Volunteers or Patients Given Concomitant Approved Interventions
Brief Title: A Study Validating the Use of Candin as a Challenge Agent in Healthy Participants - Intervention Specific Appendix 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109020; 2020-006066-37 (EudraCT Number); NOPRODPANAP1003 (Other: Janssen Research & Development, LLC); PLATFORMPANAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Candin + Tofacitinib (Experimental): Participants will receive a single dose of Candin injection on forearm of 1 arm along with a saline solution injection of 0.9 percent (%) sodium chloride (NaCl) on the opposite forearm on Day 3 and oral dose of tofacitinib for 5 days.
  Interventions: Drug: Tofacitinib
- Candin Challenge (No Intervention): All participants will receive a single dose of Candin injection on forearm of 1 arm along with a saline solution injection of 0.9% NaCl on the opposite forearm on Day 3.

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib tablet will be administered orally.
  Other Names: Xeljanz
  Arms: Candin + Tofacitinib

SUMMARY:
The purpose of this study is to characterize the delayed-type hypersensitivity (DTH) response at the site of Candin intradermal injection in the presence of a targeted immune pathway inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilograms per meter square (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of no less than 50 kilograms (kg)
* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. Any abnormalities, must be considered not clinically significant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must sign an informed consent forms (ICFs) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* A woman must agree not to donate eggs (ova, oocytes) or freeze for future use for the purposes of assisted reproduction during the study and for a period of 30 days after the last dose of study intervention

Exclusion Criteria:

* History of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic, or mucocutaneous disturbances
* History of any type of immunodeficiency or autoimmune disease or disease treatment associated with immune suppression or lymphopenia. These include but are not limited to bone marrow or organ transplantation, lymphoproliferative disorders, T- or B-cell deficiency syndromes, splenectomy, functional asplenia and chronic granulomatous disease
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Has experienced a recent single dermatomal herpes zoster eruption within the past 6 months or has had multi-dermatomal herpes zoster or central nervous system zoster within the past 5 years
* Has surgery planned within 30 days after study intervention administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Presence and Size of Induration in Active Versus Control at the Candin Injection Site Compared to the Intra-individual Saline Control Injection Site Approximately 48 Hours After Candin Challenge | Day 5
  Number of participants with presence and size of induration in active versus control at the Candin injection site compared to the intra-individual saline control injection site approximately 48 hours after Candin challenge will be reported.

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) in the Active Arm Versus the Control Arm | Up to 6 weeks
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-emergent Serious Adverse Events (SAEs) in the Active Arm Versus the Control Arm | Up to 6 weeks
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs are defined as serious events between administration of study drug and after the last dose that were absent before treatment or that worsen relative to pretreatment state.
Number of Participants with TEAEs by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) with a Frequency Threshold of 5 Percent (%) or More in the Active Arm Versus the Control Arm | Up to 6 weeks
  Number of participants with TEAEs by MedDRA SOC with a frequency threshold of 5% or more in the active arm versus the control arm will be reported. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency